CLINICAL TRIAL: NCT03957941
Title: Impact of Visual Contact With the Premature Infant on Maternal Breast Milk Expression
Brief Title: FamilyLink and Breastfeeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: 1370355
Record Dates: First submitted 2019-05-13; First posted 2019-05-21 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to the order of Intervention and Control pumping session. Excluding the first pumping session of the day, as the volume is highest at that time and more consistent throughout the rest of the day. All 30 mothers will be asked to A (Control): Pump three times while they are away from their infant without using FamilyLink for video observation of their baby during pumping and B (Intervention): Pump three times while they are away from their infant, while watching their baby via FamilyLink.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator and outcomes assessor will be blinded to the order the mothers were randomized to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FamilyLink Pumping (Experimental): Pump three times while away from infant, while watching baby via FamilyLink.
  Interventions: Behavioral: FamilyLink Pumping
- Standard Pumping (Active Comparator): Pump three times while away from infant, not watching baby via FamilyLink.
  Interventions: Behavioral: Standard Pumping

INTERVENTIONS:
Behavioral: FamilyLink Pumping — Viewing baby via FamilyLink while pumping
  Arms: FamilyLink Pumping
Behavioral: Standard Pumping — Not viewing baby via FamilyLink while pumping
  Arms: Standard Pumping

SUMMARY:
The central hypothesis guiding this project is that having mothers view live video of their babies while they are pumping increases milk volume, caloric density, and maternal pumping experience.

ELIGIBILITY:
Inclusion Criteria:

* Mothers of 30 preterm infants (born before 34 weeks gestational age) admitted to the University of California, Davis neonatal intensive care unit (NICU)
* Mother is pumping breastmilk
* Delivery at least 7 days prior
* Mother not an inpatient,

Exclusion Criteria:

* Mother has HIV
* Mother without access to a computer, smartphone, or tablet to access FamilyLink
* Infant delivered via surrogacy
* Maternal age outside limit of 18 to 50

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Mean volume of Breast Milk | Two days
  Difference in the the mean volume of breast milk expressed between intervention pumping sessions and control pumping sessions

SECONDARY OUTCOMES:
Pumping Efficiency | Three times per day for two days
  Pumping Efficiency will be calculated using the volume of breast milk expressed divided by the number of minutes of the pumping session
FamilyLink breast milk fat content | One day
  Breast milk fat content will be measured from a 5 ml sample of milk collected after a FamilyLink pumping session; The total weight and kilocalories/mL of each nutrient will be tested
Standard breast milk fat content | One day
  Breast milk fat content will be measured from a 5 ml sample of milk collected after a Standard pumping session; The total weight and kilocalories/mL of each nutrient will be tested
FamilyLink breast milk protein content | One day
  Breast milk protein content will be measured from a 5 ml sample of milk collected after a FamilyLink pumping session; The total weight and kilocalories/mL of each nutrient will be tested
Standard breast milk protein content | One day
  Breast milk protein content will be measured from a 5 ml sample of milk collected after a Standard pumping session; The total weight and kilocalories/mL of each nutrient will be tested
FamilyLink breast milk carbohydrate content | One day
  Breast milk carbohydrate content will be measured from a 5 ml sample of milk collected after a FamilyLink pumping session; The total weight and kilocalories/mL of each nutrient will be tested
Standard breast milk carbohydrate content | One day
  Breast milk carbohydrate content will be measured from a 5 ml sample of milk collected after a Standard pumping session; The total weight and kilocalories/mL of each nutrient will be tested
Quantitative pumping experience | Three times per day for two days
  Breast Milk Expression Experience Personal Experience Subscale; a five question subscale to measure participants experience with breastfeeding; the minimum score is 5 and the maximum score is 25 (higher scores indicate better outcomes)
Qualitative pumping experience | Two days
  Mothers will be asked open-ended questions, "How was your pumping experience?" "Please describe your experience watching your baby while pumping." "Would you want to use FamilyLink during pumping in the future? Why or why not?" and "Any suggestions to improve the FamilyLink pumping experience?" Responses to these items will be analyzed qualitatively.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Kair, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California-Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hoyt-Austin AE, Miller IT, Kuhn-Riordon KM, Rosenthal JL, Chantry CJ, Marcin JP, Hoffman KR, Kair LR. Bonding, Relaxation, Separation, and Connection: Expressing Human Milk While Videoconferencing with the Hospitalized Premature Infant. Breastfeed Med. 2022 Aug;17(8):653-659. doi: 10.1089/bfm.2021.0214. Epub 2022 May 23. PMID 35605051
- See also: Learn more or sign up for the study here! — https://studypages.com/s/a-study-of-the-familylink-videoconferencing-system-and-breastfeeding-305970/